CLINICAL TRIAL: NCT07178639
Title: Comparing Efficacy of Bromfenac 0.09%, Nepafenac 0.3% and Diclofenac 0.1% in Patients After Cataract Surgery
Acronym: BND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nemocnice Kolín (Other)
Responsible Party: Principal Investigator, Tomas Vanek, Study Director, Nemocnice Kolín
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025-001; 2025-001 (Other: Oblastní nemocnice Kolín a.s.)
Record Dates: First submitted 2025-07-09; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-07

CONDITIONS: Macular Oedema; Cataract Surgery; NSAID (Non-Steroidal Anti-Inflammatory Drug)
Keywords: macular oedema; cataract surgery; macular oedema treatment
MeSH Terms: conditions — Macular Edema | interventions — bromfenac; Ophthalmic Solutions; nepafenac; Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- bromfenac 0.09% (Active Comparator): Subjects will instill one drop into the study (operative) eye twice per day for a maximum of 26 days. Dosing will begin four days prior to surgery (Day 3), continue on the day of surgery and for 21 days after surgery.
  Interventions: Drug: Bromfenac 0.09 % Ophthalmic Solution
- nepafenac 0.3% (Active Comparator): Subjects will instill one drop into the study (operative) eye once per day for a maximum of 26 days. Dosing will begin four days prior to surgery (Day 3), continue on the day of surgery and for 21 days after surgery.
  Interventions: Drug: Nepafenac 0.3% Oph Susp
- diclofenac 0.1% (Active Comparator): Subjects will instill one drop into the study (operative) eye four times per day for a maximum of 26 days. Dosing will begin four days prior to surgery (Day 3), continue on the day of surgery and for 21 days after surgery.
  Interventions: Drug: diclofenac 0.1% ophthalmic susp.

INTERVENTIONS:
Drug: Bromfenac 0.09 % Ophthalmic Solution — Comparison of bromfenac ophthalmic solution 0.09% twice per day vs. nepafenac ophthalmic suspension 0.3% once per day vs. diclofenac ophthalmic suspension 0.1% four times per day for prevention of cystoid macular oedema associated with cataract surgery.
  Other Names: Bromfenac 0.09 %
  Arms: bromfenac 0.09%
Drug: Nepafenac 0.3% Oph Susp — Comparison of bromfenac ophthalmic solution 0.09% twice per day vs. nepafenac ophthalmic suspension 0.3% once per day vs. diclofenac ophthalmic suspension 0.1% four times per day for prevention of cystoid macular oedema associated with cataract surgery.
  Other Names: Nepafenac 0.3%
  Arms: nepafenac 0.3%
Drug: diclofenac 0.1% ophthalmic susp. — Comparison of bromfenac ophthalmic solution 0.09% twice per day vs. nepafenac ophthalmic suspension 0.3% once per day vs. diclofenac ophthalmic suspension 0.1% four times per day for prevention of cystoid macular oedema associated with cataract surgery.
  Other Names: diclofenac 0.1%
  Arms: diclofenac 0.1%

SUMMARY:
The goal of this clinical trial is to learn which of the drugs bromfenac 0.09%, nepafenac 0.3% and diclofenac 0.1% has better efficacy in treatment and prevention of cystoid macular oedema after cataract surgery.

The main questions it aims to answer are:

Which of the drugs has better efficacy in macular oedema prevention? What medical problems do participants have when taking different drugs? Researchers will compare drugs to each other.

Participants will:

Take on of the drugs (randomized) as their treatment in preoperative and postoperative period.

Visit the clinic after the surgery on the first day, first week, in three weeks and in six weeks.

Undergo retina examination with OCT (optical coherence tomography), best vision, and fill in forms considering their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female at least 18 years of age who require cataract surgery and no other surgical procedures during the cataract surgery.
* Agree not to have any other ocular surgical procedures in the study or fellow (non study) eye within 15 days prior to the initiation of dosing with the test article or throughout the duration of the study.
* Have a Best Corrected Visual Acuity of 20/200 or better in either eye.
* Are able to self administer test article (or have a caregiver available to instill all doses of test article).

Exclusion Criteria:

* Have known hypersensitivity to bromfenac, nepafenac, diclofenac or any component of the test article (including "procedural" medications such as anesthetic and/or fluorescein drops, dilating drops, etc.).
* Have intraocular inflammation (i.e., cells or flare in the anterior chamber as measured on slit lamp examination) in study eye at screening visit.
* Have a known blood dyscrasia or bone marrow suppression, a diagnosis of uncontrolled/unstable peptic ulcer disease, inflammatory bowel disease, or ulcerative colitis, or any uncontrolled/unstable pulmonary, cardiac, vascular, autoimmune, hepatic, renal, or central nervous system disease.
* Have used ocular, topical, or systemic NSAIDs or ocular, topical, or systemic gentamicin, or cyclosporine ophthalmic emulsion within 7 days prior to initiation of dosing with the test article or throughout the duration of study,with exception of allowing patients on a stable dose of aspirin 81 mg daily or less.
* Have diabetes of any type.
* Have any pathology of vitreoretinal interface (recognised on opcital coherence tomography).
* Have any history of pars plana vitrectomy in the study eye.
* Have glaucoma of the following types: any secondary, closed angle, severe open angle.
* Have used ocular prostaglandins within 30 days prior to initiation of dosing with test article or throughout the duration of study.
* Have active corneal pathology noted in the study eye at screening visit. Active corneal pathology is defined as corneal pathology that is non stable, or greater than mild, or will compromise assessment of the safety or efficacy of treatment. Superficial punctate keratitis in study eye.
* Have any extraocular/intraocular inflammation in the study eye at screening visit (blepharitis allowed if mild only, and no concurrent conjunctivitis or lid erythema/edema) or ongoing, unresolved uveitis.
* Have used topical, ocular, inhaled or systemic steroids within 14 days prior to screening.
* Have a history of abuse of alcohol/drugs within six months prior to the screening visit.
* Are pregnant or nursing/lactating.
* Have participated in any other study of an investigational drug or device within 30 days prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Cystoid macular oedema presence | From enrollment to the end of treatment at 6 weeks
  Measured as central retinal thickness in OCT (optical coherence tomography)

SECONDARY OUTCOMES:
Quality of life change with National Eye Institute Visual Function Questionnaire | From enrollment to the end of the treatment at 6 weeks.
  Measures the dimensions of self-reported vision-targeted health status that are most important for persons who have chronic eye diseases

CONTACTS AND LOCATIONS:
Locations (1):
- Oblastní nemocnice Kolín a.s., Kolín, Czechia

IPD SHARING:
Plan to Share IPD: No